CLINICAL TRIAL: NCT01876784
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Centre Phase III Study to Assess the Efficacy and Safety of Vandetanib (CAPRELSA™; SAR390530 (Formerly AstraZeneca ZD6474)) 300 mg in Patients With Differentiated Thyroid Cancer That Is Either Locally Advanced or Metastatic Who Are Refractory or Unsuitable for Radioiodine (RAI) Therapy
Brief Title: Evaluation of Efficacy, Safety of Vandetanib in Patients With Differentiated Thyroid Cancer
Acronym: VERIFY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D4203C00011; 2013-000422-58 (EudraCT Number); LPS14813 (Other: Sanofi)
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-06

CONDITIONS: Differentiated Thyroid Cancer
Keywords: vandetanib, AZD 6474, Differentiated Thyroid Cancer
MeSH Terms: interventions — vandetanib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vandetanib/ Vandetanib (Experimental): Participants received Vandetanib 300 mg tablet, orally once daily until disease progression or death, in randomized treatment period (up to maximum of 40 months). Participants who completed the randomized treatment period, were offered the opportunity to continue the same vandetanib treatment in the open label period, if in the investigator's opinion, they received benefit and if the participant agreed and provided their informed consent to continue the open-label period for up to additional 31 months.
  Interventions: Drug: Vandetanib (SAR390530)
- Placebo/ Vandetanib (Placebo Comparator): Participants received placebo matched to Vandetanib tablet, orally once daily until disease progression or death, in randomized treatment period (up to maximum of 40 months). Participants who completed the randomized treatment period, and experienced disease progression were offered the option of treatment in open-label period with vandetanib, if in the investigator's opinion, they received benefit and if the participant agreed and provided their informed consent to begin open-label vandetanib treatment i.e., 300 mg tablet, orally once daily for up to 31 months.
  Interventions: Drug: Vandetanib (SAR390530); Drug: Placebo

INTERVENTIONS:
Drug: Vandetanib (SAR390530) — Pharmaceutical form: tablet
  Route of administration: oral
  Other Names: CAPRELSA
Drug: Placebo — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Placebo/ Vandetanib

SUMMARY:
Primary Objective:

To determine the efficacy (as assessed by progression-free survival [PFS]) of vandetanib when compared to placebo in participants with differentiated thyroid cancer that is either locally advanced or metastatic who are refractory or unsuitable for radioiodine therapy.

Secondary Objectives:

* To determine the efficacy of vandetanib when compared to placebo in this participant population as assessed by efficacy variables including duration of response (DOR), objective response rate (ORR), change in tumour size (TS) and overall survival (OS).
* To evaluate the pharmacokinetics (PK) of vandetanib in this participant population and potentially investigate any influence of participant demography and pathophysiology on vandetanib PK.
* To demonstrate an improvement in time to worsening of pain (TWP) in participants treated with vandetanib when compared to placebo in this participant population.
* To evaluate the safety and tolerability of vandetanib treatment in this participant population.

DETAILED DESCRIPTION:
Participants who received vandetanib as randomized treatment were allowed, upon re-consent, to continue on open-label vandetanib if in the opinion of the Investigator the participant received benefit. Placebo participants who experienced disease progression within 60 days of unblinding were offered the option of treatment with open-label vandetanib if, in the Investigator's opinion, such treatment was of clinical benefit to the participant. Approximately 2 years; duration depends on individual participant response.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent to participate in the study as well as provision of informed consent to provide a sample of a previously obtained archival tumor biopsy.
* Female or male aged 18 years and older with previously confirmed histological diagnosis of locally advanced or metastatic differentiated (excluding minimally invasive follicular) thyroid cancer not amenable to surgical resection, external beam radiotherapy or local therapy.
* Measurable disease defined as at least one lesion, not irradiated within 12 weeks of the date of randomization, that can be accurately measured at baseline.
* Participants must have experienced progression within 14 months and be RAI-refractory/resistant or unsuitable for RAI.
* Thyroid-stimulating hormone (TSH) suppression below 0.5 mU/L is required.
* World Health Organization (WHO) or Eastern Cooperative Oncology Group (ECOG) Performance status 0-2.
* Negative pregnancy test (urine or serum) for female participants of childbearing potential.

Exclusion Criteria:

* Inadequate organ function as defined by: (1) Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) greater than 2.5*upper limit of normal (ULN), or greater than 5.0*ULN if judged by the Investigator to be related to liver metastases. (2) Serum bilirubin greater than 1.5*ULN. This criterion does not apply to participants with known Gilbert's Disease. (3) Creatinine clearance <50 mL/min (calculated by Cockcroft-Gault formula).
* Risk of prolonged interval between Q and T (QT) on an electrocardiogram (ECG) corrected for heart rate (QTc) as defined by: (1) Current therapy with any medication known to be associated with Torsades de pointes or potent inducers of cytochrome CYP3A4. (2) History of QT prolongation. (3) Congenital long QT syndrome. (4) QT interval corrected for heart rate by the Bazett's method (QTcB) correction unmeasurable or greater than 480 ms on screening ECG.
* Previous therapy with approved or investigational tyrosine kinase or anti- vascular endothelial growth factor (VEGF) receptor inhibitors or targeted therapies (e.g. multi-targeted kinase inhibitors such as sorafenib, AMG-706, sunitinib, pazopanib, lenvatinib).
* RAI therapy within 12 weeks prior to first dose of study drug, and radiation therapy other than RAI, including external beam, if not completed prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2013-09-17 (Actual); Primary Completion 2015-08-30 (Actual); Study Completion 2022-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (61):
- United States (10):
  - Research Site, Little Rock, Arkansas
  - Research Site, Torrance, California
  - Research Site, Lexington, Kentucky
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, New York, New York
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
- Brazil (5):
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- China (7):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Huangzhou
  - Research Site, Shanghai
  - Research Site, Tianjin
  - Research Site, Wuhan
- Czechia (2):
  - Research Site, Olomouc
  - Research Site, Prague
- Research Site, Odense, Denmark
- France (5):
  - Research Site, Angers
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Paris
  - Research Site, Villejuif
- Italy (6):
  - Research Site, Catania
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Siena
- Japan (13):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Kashiwa-shi
  - Research Site, Kobe
  - Research Site, Kōtoku
  - Research Site, Matsumoto-shi
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Shinjuku-ku
  - Research Site, Yokohama
- Poland (4):
  - Research Site, Gliwice
  - Research Site, Kielce
  - Research Site, Warsaw
  - Research Site, Zgierz
- Russia (2):
  - Research Site, Barnaul
  - Research Site, Obninsk
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, Hospitalet de Llobregat(Barcel
  - Research Site, Madrid
- Sweden (2):
  - Research Site, Lund
  - Research Site, Stockholm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 60 active centers in 12 countries. A total of 299 participants were screened between 17 September 2013 and 26 September 2014, of which 238 participants were randomized. A total of 235 participants were treated in the study.
Groups:
- Vandetanib/Vandetanib: Participants received Vandetanib 300 mg tablet, orally once daily until disease progression or death, in randomized treatment period (up to maximum of 40 months). Participants who completed the randomized treatment period, were offered the opportunity to continue the same vandetanib treatment in the open label period, if, in the investigator's opinion, they received benefit and if the participant agreed and provided their informed consent to continue the open-label period for up to additional 31 months.
- Placebo/Vandetanib: Participants received placebo matched to Vandetanib tablet, orally once daily until disease progression or death, in randomized treatment period (up to maximum of 40 months). Participants who completed the randomized treatment period, and experienced disease progression were offered the option of treatment in open-label period with vandetanib, if in the investigator's opinion, such treatment was of clinical benefit to the participant, and if the participant agreed and provided their informed consent to begin open-label vandetanib treatment i.e., 300 mg tablet, orally once daily for up to 31 months.
Period: Randomized Treatment Period (40 Months)
Arm/Group | Vandetanib/Vandetanib | Placebo/Vandetanib
Started | 119 | 119
Treated | 117 | 118
Completed | 0 | 0
Not Completed | 119 | 119
Not completed — Withdrawal by Subject | 20 | 4
Not completed — Adverse Event | 22 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — Disease progression | 43 | 81
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 1 | 0
Not completed — Development of study-specific discontinuation criteria | 5 | 2
Not completed — Randomized but not treated | 2 | 1
Not completed — Other than specified above | 24 | 25
Period: Open-label Period (31 Months)
Arm/Group | Vandetanib/Vandetanib | Placebo/Vandetanib
Started (Post completion of randomized treatment period, only eligible participants entered Open label period.) | 23 | 74
Completed | 0 | 0
Not Completed | 23 | 74
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Adverse Event | 2 | 6
Not completed — Protocol Violation | 0 | 1
Not completed — Progressive disease | 4 | 35
Not completed — Development of study-specific discontinuation criteria | 1 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 0 | 1
Not completed — Other than specified above | 9 | 18

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vandetanib/Vandetanib | Placebo/Vandetanib | Total
Number analyzed (Participants) | 119 | 119 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (9.69) | 63.2 (11.02) | 63.7 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 64 | 134
  Male | 49 | 55 | 104

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: The PFS was defined as the time (in months) from randomization until the date of first documented disease progression or death (from any cause), whichever came first. Disease progression as per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) was defined as: at least a 20% increase and absolute increase of 5 mm in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Analysis was performed by Kaplan-Meier method.
Time Frame: Randomization until disease progression or death, assessed every 12 weeks (up to 22 months)
Population: Intent to treat population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Randomized Treatment Period: Vandetanib: Vandetanib 300 mg tablet, orally once daily until disease progression or death.
- Randomized Treatment Period: Placebo: Placebo matched to vandetanib tablet, orally once daily until disease progression or death.
Arm/Group | Randomized Treatment Period: Vandetanib | Randomized Treatment Period: Placebo
Number analyzed (Participants) | 119 | 119
months | 10.0 [6.0 to 11.1] | 5.7 [5.5 to 8.4]
Statistical Analysis 1: Comparison: Randomized Treatment Period: Vandetanib vs Randomized Treatment Period: Placebo; A multiple testing procedure (MTP) with an alpha-exhaustive recycling strategy was employed to provide adequate control of type I error; Test type: Superiority or Other; p = 0.080, Log Rank — Threshold for significance at 0.05 level; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.55 to 1.03] — Vandetanib 300 mg vs Placebo

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until death due to any cause. In the absence of observation of death, survival time was censored to last date the participant is known to be alive or at the cut-off date, whichever comes first. Analysis was performed by Kaplan-Meier method.
Time Frame: From randomization to the date of death due to any cause (maximum duration: up to 42 months)
Population: Analysis was performed on intent-to-treat population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vandetanib/Vandetanib | Placebo/Vandetanib
Number analyzed (Participants) | 119 | 119
months | NA [31.6 to NA] — Median and upper limit of 95% confidence interval (CI) was not estimable due to an insufficient number of participants with events. | NA [32.1 to NA] — Median and upper limit of 95% confidence interval (CI) was not estimable due to an insufficient number of participants with events.

3. Secondary Outcome: Randomized Treatment Period: Percent Change From Baseline in Tumor Size (TS) at Week 36
Description: Tumor size was the sum of the longest diameters of the target lesions. Target lesions were measurable tumor lesions. Baseline was defined as the last evaluable assessment prior to starting treatment.
Time Frame: Baseline, Week 36
Population: Analysis was performed on intent-to-treat population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Randomized Treatment Period: Vandetanib: Participants received Vandetanib 300 mg tablet, orally once daily until disease progression or death, in randomized treatment period (up to maximum of 40 months).
- Randomized Treatment Period: Placebo: Participants received placebo matched to Vandetanib tablet, orally once daily until disease progression or death, in randomized treatment period (up to maximum of 40 months).
Arm/Group | Randomized Treatment Period: Vandetanib | Randomized Treatment Period: Placebo
Number analyzed (Participants) | 115 | 116
percent change | 23.29 (50.059) | 21.52 (25.428)

4. Secondary Outcome: Percentage of Participants With Objective Response
Description: Objective Response was defined as the percentage (%) of participants with complete response or partial response. Per RECIST 1.1 criteria, complete response was defined as the disappearance of all target lesions since Baseline. Any pathological lymph nodes selected as target lesions must have a reduction in short axis to less than (<)10 millimeters (mm). Partial response was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the Baseline sum of diameters. Progressive Disease was defined as at least at least a 20% increase and absolute increase of 5 mm in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From randomization to the date of first documented tumor progression, or death due to any cause, whichever comes first (maximum duration: up to 42 months)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Vandetanib/Vandetanib | Placebo/Vandetanib
Number analyzed (Participants) | 119 | 118
percentage of participants | 5.0 | 0

5. Secondary Outcome: Time to Worsening of Pain (TWP) Using Numeric Rating Scale (NRS) of Worst Pain
Description: Time to worsening of pain was defined as the time interval from the date of randomization to the date of first assessment of worsening of pain with no evidence of improvement within the next 14 days. Participants rate their worst pain intensity during the past seven days using an 11-point NRS scale, where 0 represents "no pain" and 10 represents "pain as bad as you can imagine." Higher scores indicated greater pain severity. TWP analysis was performed using Kaplan-Meier method.
Time Frame: From randomization to the date of first assessment of worsening of pain (maximum duration: up to 42 months)
Population: Analysis was performed on intent-to-treat population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vandetanib/Vandetanib | Placebo/Vandetanib
Number analyzed (Participants) | 119 | 119
months | 5.6 [2.9 to 8.4] | 8.3 [2.8 to 16.6]

6. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response was defined as the time from the date of first documented response until the date of documented progression or death. If participants did not progress following a response, then their DOR used the PFS censoring time. Per RECIST 1.1, progressive disease was defined as at least a 20% increase and absolute increase of 5 mm in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. DOR analysis was performed using Kaplan-Meier method.
Time Frame: From the date of first response to the date of first documented tumor progression or death due to any cause whichever comes first (maximum duration: up to 42 months)
Population: Analysis was performed on subset of participants with response. Here, '0' in 'overall number of participants' analyzed signifies that no participant in the Placebo/Vandetanib achieved any response, therefore DOR was not analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vandetanib/Vandetanib | Placebo/Vandetanib
Number analyzed (Participants) | 6 | 0
months | NA [NA to NA] — Median, upper limit and lower limit of 95%CI was not estimable due to an insufficient number of participants with events. |

7. Secondary Outcome: Randomized Treatment Period: PK Parameters: Maximum Plasma Concentration (Cmax)
Time Frame: Post-dose on Week 1 to Week 48
Population: Number of participants analyzed= participants with available data for the time points.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Randomized Treatment Period: Vandetanib
Number analyzed (Participants) | 98
ng/ml
  Week 1 | 695.1 (238.94)
  Week 2: number analyzed (Participants) | 95
  Week 2 | 846.2 (288.98)
  Week 4: number analyzed (Participants) | 93
  Week 4 | 975.7 (358.33)
  Week 8: number analyzed (Participants) | 90
  Week 8 | 1043.1 (395.08)
  Week 12: number analyzed (Participants) | 83
  Week 12 | 1041.9 (404.69)
  Week 24: number analyzed (Participants) | 61
  Week 24 | 1004.9 (408.34)
  Week 36: number analyzed (Participants) | 48
  Week 36 | 904.1 (312.51)
  Week 48: number analyzed (Participants) | 28
  Week 48 | 963.0 (452.4)

ADVERSE EVENTS:
Time Frame: The data for non-serious adverse events are presented until the Last Participant Last Visit (LPLV) date i.e., 19 June 2017, up to 3 years and 9 months. Serious adverse events were collected until the end of the study, up to 8 years and 4 months.
Description: Analysis was performed for safety population i.e., participants who received at least one dose of treatment. For participants who continued Vandetanib after the LPLV because they still benefited of it per investigator judgment, Serious adverse events were collected as long as they received treatment. No non-serious adverse events were collected after LPLV for open label period of the study.
Groups:
- Open-Label Treatment Period: Vandetanib/Vandetanib: Participants who completed the randomized treatment period, were offered the opportunity to continue the same vandetanib treatment in the open label period, if in the investigator's opinion, they received benefit and if the participant agreed and provided their informed consent to continue the open-label period for up to additional 31 months.
- Open-Label Treatment Period: Placebo/Vandetanib: Participants who completed the randomized treatment period, and experienced disease progression were offered the option of treatment in open-label period with vandetanib, if, in the investigator's opinion, such treatment was of clinical benefit to the participant, and if the participant agreed and provided their informed consent to begin open-label vandetanib treatment i.e., 300 mg tablet, orally once daily for up to 31 months.
Arm/Group | Randomized Treatment Period: Vandetanib | Randomized Treatment Period: Placebo | Open-Label Treatment Period: Vandetanib/Vandetanib | Open-Label Treatment Period: Placebo/Vandetanib
Serious Adverse Events (participants affected / at risk) | 37/117 | 19/118 | 7/23 | 24/74
Other Adverse Events (participants affected / at risk) | 111/117 | 87/118 | 9/23 | 62/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Treatment Period: Vandetanib (N=117) | Randomized Treatment Period: Placebo (N=118) | Open-Label Treatment Period: Vandetanib/Vandetanib (N=23) | Open-Label Treatment Period: Placebo/Vandetanib (N=74)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone Marrow Failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular Block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Failure Acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large Intestine Polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease Progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Impaired Healing (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple Organ Dysfunction Syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 2 (7) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 4 (4)
Post Procedural Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypobarism (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases To Spinal Cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous Cell Carcinoma Of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ivth Nerve Paresis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertebrobasilar Insufficiency (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis Noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrotic Syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (4)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 1 (1) | 1 (1)
Dermatitis Bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Henoch-Schonlein Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stevens-Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicose Vein (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Treatment Period: Vandetanib (N=117) | Randomized Treatment Period: Placebo (N=118) | Open-Label Treatment Period: Vandetanib/Vandetanib (N=23) | Open-Label Treatment Period: Placebo/Vandetanib (N=74)
Anaemia (Blood and lymphatic system disorders) | 6 (7) | 6 (8) | 1 (1) | 0 (0)
Cornea Verticillata (Eye disorders) | 9 (9) | 0 (0) | 1 (1) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 8 (9) | 8 (9) | 0 (0) | 3 (3)
Abdominal Pain Upper (Gastrointestinal disorders) | 6 (9) | 4 (4) | 1 (1) | 6 (6)
Constipation (Gastrointestinal disorders) | 9 (11) | 11 (13) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 77 (126) | 24 (29) | 3 (5) | 39 (58)
Dry Mouth (Gastrointestinal disorders) | 6 (6) | 2 (2) | 1 (1) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 6 (7) | 3 (4) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 22 (24) | 17 (21) | 1 (1) | 16 (20)
Stomatitis (Gastrointestinal disorders) | 6 (6) | 3 (3) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 9 (14) | 12 (15) | 1 (1) | 6 (7)
Asthenia (General disorders) | 21 (27) | 15 (15) | 1 (1) | 7 (8)
Fatigue (General disorders) | 13 (14) | 13 (13) | 1 (1) | 14 (14)
Non-Cardiac Chest Pain (General disorders) | 3 (3) | 0 (0) | 0 (0) | 5 (6)
Pyrexia (General disorders) | 6 (7) | 10 (14) | 0 (0) | 6 (6)
Hepatic Function Abnormal (Hepatobiliary disorders) | 6 (7) | 0 (0) | 0 (0) | 3 (3)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Nasopharyngitis (Infections and infestations) | 8 (10) | 7 (9) | 0 (0) | 3 (3)
Paronychia (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 4 (4)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (5) | 7 (8) | 0 (0) | 1 (2)
Urinary Tract Infection (Infections and infestations) | 11 (16) | 3 (4) | 0 (0) | 4 (5)
Alanine Aminotransferase Increased (Investigations) | 16 (23) | 4 (6) | 0 (0) | 12 (13)
Aspartate Aminotransferase Increased (Investigations) | 15 (21) | 4 (7) | 0 (0) | 8 (10)
Blood Creatinine Increased (Investigations) | 7 (9) | 1 (1) | 0 (0) | 6 (6)
Electrocardiogram Qt Prolonged (Investigations) | 36 (55) | 4 (6) | 1 (1) | 20 (36)
Weight Decreased (Investigations) | 10 (11) | 3 (4) | 0 (0) | 7 (8)
Decreased Appetite (Metabolism and nutrition disorders) | 21 (23) | 2 (2) | 1 (1) | 15 (19)
Hypocalcaemia (Metabolism and nutrition disorders) | 17 (18) | 3 (3) | 1 (1) | 6 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (11) | 5 (5) | 0 (0) | 7 (11)
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 (19) | 1 (1) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (11) | 5 (5) | 0 (0) | 4 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 12 (14) | 2 (2) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 9 (9) | 0 (0) | 6 (7)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 10 (11) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 16 (23) | 9 (11) | 0 (0) | 7 (10)
Anxiety (Psychiatric disorders) | 6 (6) | 5 (5) | 0 (0) | 4 (4)
Insomnia (Psychiatric disorders) | 15 (15) | 2 (2) | 0 (0) | 10 (11)
Haematuria (Renal and urinary disorders) | 7 (7) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 8 (8) | 0 (0) | 1 (1) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 12 (16) | 1 (1) | 12 (14)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 0 (0) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 10 (10) | 0 (0) | 7 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 8 (9) | 0 (0) | 3 (3)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (7) | 0 (0) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 9 (9) | 2 (2) | 0 (0) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (3) | 0 (0) | 1 (1)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 13 (14) | 2 (2) | 0 (0) | 6 (9)
Dry Skin (Skin and subcutaneous tissue disorders) | 18 (18) | 6 (6) | 0 (0) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 5 (7) | 2 (2) | 0 (0) | 6 (7)
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 6 (7) | 0 (0) | 0 (0) | 5 (5)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 14 (15) | 0 (0) | 0 (0) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5) | 1 (1) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 36 (51) | 6 (7) | 0 (0) | 19 (24)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1) | 0 (0) | 3 (5)
Hypertension (Vascular disorders) | 48 (53) | 9 (9) | 0 (0) | 31 (35)

LIMITATIONS AND CAVEATS:
This study was part of the drug acquisition where model-based PK analysis was not performed by the legacy company. Available PK descriptive statistics have been reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.